CLINICAL TRIAL: NCT03456258
Title: Lactoferrin Versus Ferrous Sulphate for the Treatment of Iron Deficiency Anemia During Pregnancy,a Randomized Clinical Trial
Brief Title: Lactoferrin Versus Ferrous Sulphate for the Treatment of Iron Deficiency Anemia During Pregnancy
Acronym: Lactoferrin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Ragab, Principal investigator, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ainshams maternity hospital
Record Dates: First submitted 2018-02-23; First posted 2018-03-07 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Iron Deficiency Anemia of Pregnancy
MeSH Terms: interventions — Blood Cell Count

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactoferrin (Experimental): To measure hemoglobin difference and serum ferritin
  Interventions: Diagnostic Test: Complete blood count
- Ferrous sulphate (Experimental): To measure hemoglobin difference and serum ferritin
  Interventions: Diagnostic Test: Complete blood count

INTERVENTIONS:
Diagnostic Test: Complete blood count — To measure hemoglobin difference and serum ferritin levels .
  Other Names: Serum ferritin

SUMMARY:
The study aims to compare the efficacy and the safety of Lactoferrin versus ferrous sulphate for the treatment of iron deficiency anemia during pregnancy.

DETAILED DESCRIPTION:
The study was done at ainshams university maternity hospital on 100 pregnant women randomized in two groups .

Group one lactoferrin group Group two ferrous sulphate group

ELIGIBILITY:
Inclusion Criteria:

* pregnant women from 20 to 40 years
* iron deficiency anemia (mild and moderate)
* gestational age 13 to 26 weeks
* singleton viable pregnancy.

Exclusion Criteria:

* history of anemia due to chronic blood loss
* hemolytic anemia
* severe anemia
* history of peptic ulcer

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
hemoglobin level | 2 months
  Measure hemoglobin level two months after treatment

SECONDARY OUTCOMES:
Serum ferritin | 2 months
  Measure serum ferritin level

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Ragab, MBBCH, Principal Investigator — Ainshams university maternity hospital
Locations (1):
- Ainshams maternity hospital, Cairo, Abbasia, Egypt